CLINICAL TRIAL: NCT00001522
Title: Population Differences in the Insulin Sensitivity, Resting Energy Expenditure, and Body Composition of Overweight Children and Children of Overweight Parents
Brief Title: Metabolic Differences of Overweight Children and Children of Overweight Parents
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 960101; 96-CH-0101
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2019-09-23 (Actual); Status verified 2018-04-12

CONDITIONS: Obesity
Keywords: Insulin Resistance; Race; Body Fat; Body Composition; Obesity
MeSH Terms: conditions — Obesity; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study focuses on the way weight is gained. Individuals who gain weight primarily in their midsection (visceral weight) are at an increased risk for developing diabetes and high blood pressure.

Research has shown that African Americans suffer more often from high blood pressure, diabetes (non-insulin dependent), and heart disease than Caucasian Americans. These conditions lead to significant numbers of deaths and diseases associated with and made worse by obesity.

African American women in particular suffer from obesity and the associated conditions of obesity more than any other race or gender. However, it is unknown if the conditions seen in African American women are a result of the obesity or differences in their insulin sensitivity, glucose disposal, or fat metabolism.

This study will compare body composition, total and resting energy expenditure, and glucose disposal of obese African American and Caucasian children and of non-obese children of obese African American and Caucasian parents, to characterize the timing and nature of factors that may contribute to the prevalence of obesity and its complications.

Patients participating in this study will be followed for 15 years and be evaluated every 5 years during the study.<TAB>

DETAILED DESCRIPTION:
African Americans have a greater prevalence than Caucasian Americans of hypertension, non-insulin-dependent diabetes mellitus, and cardiovascular disease. These conditions lead to substantial excess morbidity and mortality and are associated with and exacerbated by obesity, the prevalence of which is strikingly elevated in African American women. It is unknown if this increased prevalence of comorbid conditions is solely related to the greater prevalence of severe obesity among African American women, or due to differences in insulin sensitivity, glucose disposal, body composition, or fat cell metabolism. Through this project, we have verified that many of the physiological differences observed between African American and Caucasian adults are already present in obese children and in children at high risk for developing obesity. However, the roles that differences in energy expenditure, glucose metabolism, body composition, and other factors play in determining which children develop obesity and its comorbid conditions in adulthood remain unclear. In this study, we compare body composition, total and resting energy expenditure, and glucose disposal of obese African American and Caucasian children and of non-obese children of obese African American and Caucasian parents, to characterize the timing and nature of factors that may contribute to the prevalence of obesity and its complications. We also relate serum levels of the body-fat related circulating factors such as leptin, to these measures, and obtain samples for genomic DNA isolation from participants and their parents to characterize the roles of genes felt important for the development of obesity. We will follow these children for 15 years, studying them intensively at 5 year intervals until adulthood.

ELIGIBILITY:
* INCLUSION CRITERIA:

Volunteers will qualify for inclusion under this protocol if they meet the following criteria:

1. Good general health. Individuals with renal, hepatic, most endocrinologic (e.g. hypothyroidism, or Cushing syndrome), or pulmonary disorders (other than mild asthma not requiring chronic medication) will be excluded.
2. For obese subjects, body mass index for age above the 85th percentile (determined by NHANES I age-, sex-, and race-special data). For normal weight subjects of obese parents, body mass index (determined by NHANES I age-, sex-, and race- specific data) between the 5th and 85th percentile and both parents' current body mass index above 25 kg/m(2), or a history of a body mass index above 25 kg/m(2).
3. No significant psychiatric illness.
4. At initial visit, Tanner I (prepubertal) or Tanner II (early pubertal) pubic hair and breast stage of development for girls, and Tanner I or Tanner II pubic hair and testes size (6ml) for boys.
5. Subjects must be able to undergo MRI. Volunteers with metal in their bodies that are contraindications for MRI will be excluded. These include cardiac pacemakers, neural pacemakers, aneurysmal clips, shrapnel, ocular foreign bodies, cochlear implants, non-detachable electronic or electromechanical devices (such as infusion pumps, nerve stimulators, bone growth stimulators, etc.).
6. Age 6 to12 years at the start of the study.
7. For girls who have been followed to an age when they are menstruating (or are of an age when pregnancy is a possibility), a negative pregnancy test.
8. Race of all 4 grandparents self-identified either as all Caucasian or all African American.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 1996-06-06; Study Completion 2018-04-12

PRIMARY OUTCOMES:
Adiposity | Yearly for 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Jack A Yanovski, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Yanovski SZ, Reynolds JC, Boyle AJ, Yanovski JA. Resting metabolic rate in African-American and Caucasian girls. Obes Res. 1997 Jul;5(4):321-5. doi: 10.1002/j.1550-8528.1997.tb00558.x. PMID 9285838
- [Background] Yanovski JA, Yanovski SZ, Gold PW, Chrousos GP. Differences in the hypothalamic-pituitary-adrenal axis of black and white women. J Clin Endocrinol Metab. 1993 Aug;77(2):536-41. doi: 10.1210/jcem.77.2.8393890.
- [Background] Ravussin E. Energy metabolism in obesity. Studies in the Pima Indians. Diabetes Care. 1993 Jan;16(1):232-8. doi: 10.2337/diacare.16.1.232. PMID 8422781
- [Derived] Omotosho YB, Reynolds JC, Yanovski JA, Tatsi C. Body Composition and Fat Deposition in Children with Cushing Disease and Associations with Cardiometabolic Risk Factors. J Pediatr. 2025 Dec 3;290:114933. doi: 10.1016/j.jpeds.2025.114933. Online ahead of print. PMID 41349930
- [Derived] Manoli I, Sysol JR, Head PE, Epping MW, Gavrilova O, Crocker MK, Sloan JL, Koutsoukos SA, Wang C, Ktena YP, Mendelson S, Pass AR, Zerfas PM, Hoffmann V, Vernon HJ, Fletcher LA, Reynolds JC, Tsokos MG, Stratakis CA, Voss SD, Chen KY, Brown RJ, Hamosh A, Berry GT, Chen XS, Yanovski JA, Venditti CP. Lipodystrophy in methylmalonic acidemia associated with elevated FGF21 and abnormal methylmalonylation. JCI Insight. 2024 Feb 22;9(4):e174097. doi: 10.1172/jci.insight.174097. PMID 38271099
- [Derived] Ballenger KL, Tugarinov N, Talvacchio SK, Knue MM, Dang Do AN, Ahlman MA, Reynolds JC, Yanovski JA, Marini JC. Osteogenesis Imperfecta: The Impact of Genotype and Clinical Phenotype on Adiposity and Resting Energy Expenditure. J Clin Endocrinol Metab. 2022 Jan 1;107(1):67-76. doi: 10.1210/clinem/dgab679. PMID 34519823
- [Derived] Demidowich AP, Parikh VJ, Dedhia N, Branham RE, Madi SA, Marwitz SE, Roberson RB, Uhlman AJ, Levi NJ, Mi SJ, Jun JY, Broadney MM, Brady SM, Yanovski JA. Associations of the melanocortin 3 receptor C17A + G241A haplotype with body composition and inflammation in African-American adults. Ann Hum Genet. 2019 Sep;83(5):355-360. doi: 10.1111/ahg.12315. Epub 2019 Apr 2. PMID 30937899
- [Derived] Han JC, Reyes-Capo DP, Liu CY, Reynolds JC, Turkbey E, Turkbey IB, Bryant J, Marshall JD, Naggert JK, Gahl WA, Yanovski JA, Gunay-Aygun M. Comprehensive Endocrine-Metabolic Evaluation of Patients With Alstrom Syndrome Compared With BMI-Matched Controls. J Clin Endocrinol Metab. 2018 Jul 1;103(7):2707-2719. doi: 10.1210/jc.2018-00496. PMID 29718281
- [Derived] Radin RM, Tanofsky-Kraff M, Shomaker LB, Kelly NR, Pickworth CK, Shank LM, Altschul AM, Brady SM, Demidowich AP, Yanovski SZ, Hubbard VS, Yanovski JA. Metabolic characteristics of youth with loss of control eating. Eat Behav. 2015 Dec;19:86-9. doi: 10.1016/j.eatbeh.2015.07.002. Epub 2015 Jul 18. PMID 26210388
- [Derived] Tanofsky-Kraff M, Shomaker LB, Stern EA, Miller R, Sebring N, Dellavalle D, Yanovski SZ, Hubbard VS, Yanovski JA. Children's binge eating and development of metabolic syndrome. Int J Obes (Lond). 2012 Jul;36(7):956-62. doi: 10.1038/ijo.2011.259. Epub 2012 Jan 10. PMID 22234282
- [Derived] Shomaker LB, Tanofsky-Kraff M, Stern EA, Miller R, Zocca JM, Field SE, Yanovski SZ, Hubbard VS, Yanovski JA. Longitudinal study of depressive symptoms and progression of insulin resistance in youth at risk for adult obesity. Diabetes Care. 2011 Nov;34(11):2458-63. doi: 10.2337/dc11-1131. Epub 2011 Sep 12. PMID 21911779